CLINICAL TRIAL: NCT00088855
Title: Phase II Study of Bortezomib (PS-341) and Pegylated Liposomal Doxorubicin as Initial Therapy for Adult Patients With Symptomatic Multiple Myeloma
Brief Title: Bortezomib and Pegylated Liposomal Doxorubicin Hydrochloride in Treating Patients With Previously Untreated Symptomatic Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01607; NCI-2014-01607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2012-02810; CDR377483; CALGB 10301 (Other: Alliance for Clinical Trials in Oncology); CALGB-10301 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma
MeSH Terms: interventions — Bortezomib; liposomal doxorubicin; Doxorubicin

ARMS (1):
- Treatment (bortezomib and pegylated liposomal doxorubicin) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 4. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Other: Laboratory Biomarker Analysis; Drug: Pegylated Liposomal Doxorubicin Hydrochloride

INTERVENTIONS:
Drug: Bortezomib — Given IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pegylated Liposomal Doxorubicin Hydrochloride — Given IV
  Other Names: ATI-0918; Caelyx; DOX-SL; Doxil; Doxilen; Doxorubicin HCl Liposomal; Doxorubicin HCl Liposome; doxorubicin hydrochloride liposome; Duomeisu; Evacet; LipoDox; Lipodox 50; Liposomal Adriamycin; liposomal doxorubicin hydrochloride; Liposomal-Encapsulated Doxorubicin; Pegylated Doxorubicin HCl Liposome; S-Liposomal Doxorubicin; Stealth Liposomal Doxorubicin; TLC D-99

SUMMARY:
This phase II trial studies the side effects and how well bortezomib and pegylated liposomal doxorubicin hydrochloride work in treating patients multiple myeloma that are experiencing symptoms and have not received prior treatment. Bortezomib and pegylated liposomal doxorubicin hydrochloride may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the complete response (CR) + near-complete response (nCR) rate of the bortezomib/pegylated liposomal doxorubicin (pegylated liposomal doxorubicin hydrochloride) regimen in patients with previously untreated, symptomatic multiple myeloma.

II. To evaluate the toxicity of the bortezomib/pegylated liposomal doxorubicin regimen in patients with previously untreated, symptomatic multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate, including patients with CR, nCR, and partial response (PR), of the bortezomib/pegylated liposomal doxorubicin regimen in patients with previously untreated, symptomatic multiple myeloma.

II. To evaluate the impact of therapy with the bortezomib/pegylated liposomal doxorubicin regimen on the ability to collect peripheral blood stem cells in those patients going on to subsequent autologous stem cell transplantation.

III. To evaluate the time to progression (TTP) in all patients receiving bortezomib/pegylated liposomal doxorubicin therapy, both those who go on to autologous stem cell transplantation and those who do not go on to transplantation.

IV. To evaluate the value of early changes in levels of serum interleukin 6 (IL-6) and macrophage inflammatory protein 1 alpha (MIP-1α) as predictors of response to bortezomib/pegylated liposomal doxorubicin.

V. To correlate pre-treatment clinical and biological characteristics with response to therapy and toxicity.

OUTLINE:

Patients receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11 and pegylated liposomal doxorubicin hydrochloride IV over 1 hour on day 4. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 weeks for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of symptomatic multiple myeloma with evaluable disease parameters
* A diagnosis of symptomatic multiple myeloma requires:

  * A monoclonal serum and/or urine protein
  * Clonal bone marrow plasmacytosis, or a histologically confirmed plasmacytoma
  * Related organ or tissue impairment, consisting of:

    * Hypercalcemia (serum calcium > 0.25 mmol/l above the upper limit of normal, or > 2.75 mmol/l [i.e. > 11.5 mg/dl]) AND/OR
    * Renal insufficiency (serum creatinine > 173 mmol/l [i.e., > 2 mg/dL]); (please note that serum creatinine may not be >= 2.5 mg/dL) AND/OR
    * Anemia (hemoglobin 2 g/dl below the lower limit of normal, or hemoglobin < 10 g/dl) AND/OR
    * Bony lesions (lytic bony lesions, or osteoporosis with compression fractures) AND/OR
    * Other findings, such as symptomatic hyperviscosity, amyloidosis, or recurring bacterial infections (> 2 episodes in 12 months)
* Patients may not have undergone any prior therapy, with the following exceptions:

  * Prior plasmapheresis with plasma exchange (PLEX) for a hyperviscosity syndrome is allowed, providing the patient has no current evidence of hyperviscosity and has not required PLEX for at least one week prior to initiation of therapy
  * Prior radiation therapy to areas of spinal cord compression by plasmacytomas, painful lesions due to bony involvement, or other myeloma-related indications, is allowed provided that radiation will have been completed 3 weeks before initiation of therapy
  * Prior surgical intervention, such as for bony fractures or other myeloma-related complications, is allowed provided that this will have been completed 3 weeks before the initiation of therapy, and patients have recovered from surgery
  * Prior therapy with corticosteroids for indications other than multiple myeloma is allowed, provided such therapy has been discontinued at least two weeks prior to study entry, and at least two weeks before their baseline disease evaluation
  * Prior supportive therapy with bisphosphonates or erythropoietin is allowed
* Inclusion of females of childbearing potential requires a negative pregnancy test
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients may not have a prior history of a hypersensitivity reaction to pegylated liposomal doxorubicin or doxorubicin, bortezomib or other boronic acid-based compounds

  * Patients with a history of reactions to liposomal drug formulations other than pegylated liposomal doxorubicin will be evaluated individually, and if their reactions were felt to have been due to the liposomal component itself, as opposed to the encapsulated agent, they will be excluded at the discretion of the investigators
* Patients who are known to be human immunodeficiency virus (HIV)-seropositive and are taking anti-retrovirals may not participate in this study; patients who are HIV-seropositive and not on anti-retroviral therapy, and who otherwise meet the organ function criteria, will be eligible for the study
* Patients who are known to have active hepatitis A, B, or C viral infection may not participate in this study
* No electrocardiogram (EKG) evidence of acute ischemia
* No EKG evidence of medically significant conduction system abnormalities
* No history of myocardial infarction within the last 6 months
* Left ventricular ejection fraction (LVEF) must be >= 45% by either echocardiography or radionuclide-based multiple gated acquisition (radionuclide ventriculography [RNV] or multiple gate acquisition scan [MUGA])
* No class 3 or class 4 New York Heart Association congestive heart failure
* Creatinine < 2.5 mg/dL
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) and aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 times the upper limit of the institutional normal value
* Total bilirubin =< 1.2 times the upper limit of the institutional normal value
* Absolute neutrophil count (ANC) >= 1,000/ul
* Platelets >= 100,000/ul
* Hemoglobin >= 8 g/dl (transfusion- and/or growth factor-dependent patients are not excluded if the above parameters can be achieved with such support)
* For those patients receiving warfarin (Coumadin), unfractionated heparin, or low-molecular weight heparin therapy, the applicable coagulation parameter that is being monitored must be within the accepted therapeutic ranges for those indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-06-15 (Actual); Primary Completion 2006-10-31 (Actual); Study Completion 2008-01-08 (Actual)

PRIMARY OUTCOMES:
CR+nCR rate | After 18 weeks (6 courses of treatment)
  Will be estimated with an exact 90% confidence interval.

SECONDARY OUTCOMES:
CR+nCR+PR rate | After 18 weeks (6 courses of treatment)
  Will be estimated with an exact 90% confidence interval.
Maximal response rate | After 18 weeks (6 courses of treatment)
Incidence of adverse events, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 5 years
  Toxicities will be tabulated by type and grade.
Progression-free survival | From on-study date to the date of progression or death, whichever comes first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Overall survival | From on-study date to the date of death, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Changes in IL-6 and MIP-1 | Baseline to up to day 2 of course 1
  The association of response with pre-treatment characteristics such as cytogenetics and fluorescence in situ hybridization and with early changes in IL-6 and MIP-1 will be described by reporting response rates (and their confidence intervals) according to subgroup (e.g., response rates by age group; response rates by large/small change in IL-6 level).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Z Orlowski, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (25):
- United States (25):
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Frisbie Hospital, Rochester, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Lenoir Memorial Hospital, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia